CLINICAL TRIAL: NCT06979193
Title: Effectiveness of Peer Counseling in Addressing Psychological Distress and Exposure to Violence Among LGBTIQA+ Population in Nepal: A Three-arm Randomized Controlled Trial
Brief Title: Peer Counselling to Reduce Psychological Distress and Exposure to Violence Among Sexual and Gender Minorities
Acronym: SAATHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Public Health and Environment Research Centre (PERC), Nepal (Other)
Collaborators: Department of Global Public Health and Primary Care, University of Bergen (Unknown); Blue Diamond Society, Nepal (Unknown); Sahayatri Samaj, Parsa (Unknown); Friends Hetauda, Makwanpur (Unknown); Pahichan Nepal, Sarlahi (Unknown); Manab Sachet Samaj, Chitwan (Unknown); Sunaulo Bihani Samaj, Dhanusha (Unknown); CruiseAIDS Nepal, Kathmandu (Unknown); Parichaya Samaj, Lalitpur (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 398_2024
Record Dates: First submitted 2025-05-12; First posted 2025-05-18 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Mental Health; Psychological Distress; Secondary Violence Reduction; Discrimination; Sexual and Gender Minorities; Minority Groups; Homosexuality; Domestic Violence; Gender Based Violence
Keywords: Problem Management Plus; LGBTIQA+; Mental Health Services; RCT; Nepal; Peer Counseling; Violence Prevention; Psychological Support; Participatory Research
MeSH Terms: conditions — Psychological Well-Being; Coitus; Homosexuality

STUDY DESIGN:
Intervention Model Description: Study participants will be randomly assigned to one of the three arms. The control arm (Arm 1) will receive standard care, whereas the second intervention arm (Arm 2) will receive six weekly counselling sessions (approximately 90 minutes each) on Problem Management Plus strategies, safety planning, and empowerment-based counselling. The third intervention arm (Arm 3) will receive the same counseling as Arm 2, along with 11 additional monthly group meetings to enhance social support. Participants will be followed for one year to assess the outcomes of interest.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors will be independent from the intervention team and will not be involved in delivering the intervention. They will be masked to participant's group assignment in order to reduce bias, ensure objective data collection, and minimize measurement bias during the assessment of study outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Arm (Arm 1)- Usual Standard Care (No Intervention): Standard care includes all available mental health and violence prevention services in the study area. If participants are found to have severe psychological distress or are at risk of suicide at any time during the study, they will be referred to a mental health professional. The study team includes psychiatrists and psychosocial counselors who will be available to provide remote counseling or in-person consultations, if needed. If free services are not available, the study will arrange appointments, cover consultation fees, and support travel costs for up to five sessions. A leaflet with mental health information, practical tips, and contact details for support organizations (including 24-hour suicide prevention hotlines) will be provided. Participants will also be referred to One Stop Crisis Management Centers for counseling, medical treatment, and legal support for survivors of violence.
- Arm 2- SAATHI intervention (Augmented PM+ counseling) (Experimental): In addition to standard care, participants in the SAATHI intervention (Arm 2) will receive peer-led augmented Problem Management Plus (PM+) counseling, along with safety planning.
  Interventions: Behavioral: SAATHI intervention (Augmented PM+ counseling)
- Arm 3- SAATHI intervention with Peer-Led Group Meetings (Experimental): Participants in Intervention Arm 3 will receive the same counselling as those in Arm 2, consisting of six weekly peer-led sessions. In addition, they will take part in 11 monthly peer-led group support meetings.
  Interventions: Behavioral: SAATHI intervention with Peer-Led Group Meetings

INTERVENTIONS:
Behavioral: SAATHI intervention (Augmented PM+ counseling) — Study participants in this arm will attend six weekly peer-led sessions, each approximately 90-minutes in length, designed to empower them to make decisions about their lives and build resilience. PM+ is a psychological intervention developed by the World Health Organization, based on principles of cognitive behavioural therapy. It includes components such as understanding adversity and psychoeducation on mental health, managing stress, problem-solving, behavioural activation, and strengthening social support. The PM+ model in this study is augmented with additional elements, including self-empowerment strategies, motivational interviewing, psychoeducation on intimate partner and community violence, mindful meditation and safety planning. Participants will also be introduced to best practices and lessons learned that support danger assessments and avoidance of risk of future violence. The intervention aims to improve participants' overall circumstances and mental well-being.
  Arms: Arm 2- SAATHI intervention (Augmented PM+ counseling)
Behavioral: SAATHI intervention with Peer-Led Group Meetings — These 11-monthly peer-led group sessions are designed to enhance social support, build resilience, and reinforce the application of augmented PM+ strategies in daily life. They provide a safe space for reflection and mutual encouragement among study participants. The group sessions focus on managing stress, strengthening self-regulation, building self-esteem, fostering social connectedness, and promoting positive identity development.
  Group sessions involve identifying and discussing the barriers and facilitators related to practicing slow breathing techniques, problem-solving strategies, maintaining physical activity, navigating intimate partner and community violence, understanding social support networks, and planning for safety in various situations faced by sexual and gender minorities.
  Arms: Arm 3- SAATHI intervention with Peer-Led Group Meetings

SUMMARY:
Lesbian, Gay, Bisexual, Transgender, Intersex, Queer, Asexual, and other sexually or gender diverse (LGBTIQA+) communities in many countries face high levels of mental health problems compared to the general population. This is often due to discrimination, being excluded, abuse, and unfair treatment. In many low- and middle-income countries, including Nepal, the mental health needs of LGBTIQA+ people are not met, and the violence they experience is often ignored because they are seen as breaking gender norms. The low number of trained mental health specialists in a country like Nepal imply that any short-term effort to alleviate the mental health problems among LGBTIQA+ must rely on other type of support workers such as peers. There is growing evidence that help from community members-such as counselling given by non-professionals-can improve mental well-being. Considering that discrimination of LGBTIQA+ is common also within the health services, this study will look at whether peer counselling-support provided by trained LGBTIQA+ community members-can work well in Nepal. We have improved a counselling program called 'Problem Management Plus' (PM+), developed by the World Health Organization, by adding new parts that focus on reducing the risk of some of the contributing causes of mental distress, namely violence, marginalisation and loneliness. The added components include safety planning, counselling that builds confidence and strength, and goal setting strategies to help study participants use the skills they learn and reach the desired impact. In addition, peer-led monthly group meetings will be conducted to enhance social cohesion, strengthen interpersonal networks, and reduce feeling of loneliness. The study uses a community based participatory research approach, meaning LGBTIQA+ people are invited to give inputs throughout the study from study design to being involved as peer advocates to deliver the counselling. The trial will recruit at least 960 LGBTIQA+ individuals aged 18 to 55 years living in seven districts of Nepal. Study participants will be randomly allocated to one of three arms: one arm receiving individual augmented PM+ counselling with six weekly sessions; one arm receiving the individual augmented PM+ counselling followed by 11 monthly group sessions; and one control arm. There will be a one year follow-up to examine whether the peer support helps improve mental health and reduce exposure to violence among LGBTIQA+ people. The study findings will help guide programmes to improve the mental health of LGBTIQA+ in other low- and middle-income countries where they also experience discrimination, exclusion, and violence.

DETAILED DESCRIPTION:
Sexual and gender minorities, including Lesbian, Gay, Bisexual, Transgender, Intersex, Queer, Asexual and other sexually or gender diverse (LGBTIQA+) individuals, disproportionately experience social stressors such as discriminatory attitudes, violence, prejudice, and stigmatization. This environment leads to negative health outcomes, including physical ailments and risky health-related behaviors (e.g., smoking, drug abuse, and inconsistent condom usage), as well as mental health problems, ultimately impacting the overall well-being of these vulnerable groups. LGBTIQA+ individuals often anticipate rejection and discrimination from the majority population, which leads to constant vigilance, identity concealment, and self-stigma. These factors negatively affect self-acceptance and exacerbate psychological distress. Despite the high burden of violence and mental illness, LGBTIQA+ individuals tend to use health services less frequently than the majority population in many countries. This is due to fears of discrimination also from health professionals and prior experiences of disrespectful treatment and poor communication. To meet the violence prevention and mental health needs of LGBTIQA+ individuals in low- and middle-income countries (LMICs) and reduce health inequalities, culturally relevant, low-cost interventions that do not require highly trained professionals are needed.

The overall objective of this trial is to evaluate the effectiveness of a multicomponent intervention (SAATHI) in reducing exposure to violence and psychological distress among LGBTIQA+ people in Nepal. This project utilizes a mixed-method research design, and the trial had been preceded by formative research with qualitative interviews and focus group discussions with key stakeholders to evaluate the feasibility and acceptability of the intervention package. The three-armed randomized controlled trial will be implemented in seven districts across two provinces in Nepal. A qualitative process evaluation will be conducted during the intervention delivery.

We will enroll at least 960 LGBTIQA+ participants in the trial. The inclusion criteria are: age 18-55 years, history of surviving violence in the previous 12 months, and a score of ≥3 on the General Health Questionnaire indicating psychological distress.

The participants allocated to the two intervention arms will receive six weekly 90-minute counseling sessions covering multiple topics. The counselling aims to mitigate the psychological effects of trauma and moderate the impacts of a stressful, coercive, and threatening environment by altering individuals' appraisal of stressful events, modify coping patterns, and promote self-regulation, self-esteem, and positive feelings about LGBTIQA+ identity. In one of the intervention arms the participants will also be invited to 11 monthly group sessions after the individual counselling to enhance social support and social cohesiveness. The counselling and the group sessions will be offered by peer advocates who have received a 10-day training in counselling and group facilitation.

The trial participants will be followed up for one year to assess changes in exposure to violence and mental health status. The primary outcome will be GHQ-12 score. The effectiveness analysis will be based on intention-to-treat principles. The intervention effects on outcomes will be assessed using mean differences for continuous outcomes and risk ratios and absolute risk differences for binary variables.

The qualitative analysis of data from the formative research and intervention delivery will be based on Reflexive Thematic Analysis, grounded in critical realist/contextualist ontology, where interviewees' experiences are understood as lived realities produced and existing within broader social contexts.

By addressing mental health distress, discrimination and violence through a culturally sensitive and community-driven approach, this study aims to contribute to the reduction of health disparities and the improvement of health and well-being among LGBTIQA+ individuals in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as a member of the LGBTIQA+ community
* Aged 18 to 55 years
* Have a history of exposure to any form of violence (physical, sexual, or psychological) within the past 12 months
* Exhibit psychological distress, defined as a score of more than or equal to 3 on the General Health Questionnaire (GHQ-12)

Exclusion Criteria:

* Express current suicidal ideation or plans to end their life
* Meet diagnostic criteria for substance use disorders, including alcohol or drug dependence
* Have severe functional impairment due to a mental, neurological, or developmental disorder (e.g., severe intellectual disability, dementia, or psychosis)
* Decline or are unable to provide informed consent
* Intend to relocate from the study districts or move outside the country within the next few months

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 960 (Estimated)
Dates: Start 2025-05-20 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
General Health Questionnaire (GHQ-12) | Baseline Assessment; Follow up at 47 weeks after SAATHI counselling completion (53 weeks after baseline assessment). Note: This variable will also be assessed as a secondary outcome at 7 weeks and 18 weeks after baseline.
  The General Health Questionnaire (GHQ-12) will be used to assess psychological distress among study participants. The GHQ-12 consists of 12-items and, when scored using the Likert method, resulting in a total score ranging from 0 to 36, with higher scores indicate greater levels of psychological distress. Participants will be asked to reflect on their experiences over the past two weeks. The mean score will be used as a measure of mental distress.
Experience of violence | Baseline Assessment; Follow up at 53 weeks after baseline assessment. Note: Experiences of violence (type-specific violence and severity/high-intensity violence) as a secondary outcome will be assessed at 18 weeks and at 12 months.
  Experience of violence will be measured using a modified version of WHO multi-country questionnaire on women's health and domestic violence. The adapted tool assesses the prevalence and type of violence experienced by study participants at different time points. This will be measured as a binary variable with the value 1 if a participant has experienced any type of violence in the specified recall period, and 0 if they have not experienced any recent violence.
  The following categories are included in the definition of violence: controlling behaviors, psychological violence, physical violence, and sexual violence. The recall period for experience of violence at baseline will be the past 12 months. Changes in the experience of violence at follow-up assessments will be measured relative to baseline.

SECONDARY OUTCOMES:
Post-Traumatic Stress Disorder Symptoms (PCL-5) | Baseline Assessment; Follow up at one-week post-counselling (7 weeks after baseline); Follow up at 47 weeks post-counselling (53 weeks after baseline)
  Post-Traumatic Stress Disorder (PTSD) Symptoms will be measured using PTSD checklist for DSM-5 (PCL-5), which is a 20-item self-report measure used to assess the presence and severity of PTSD in the previous week, based on DSM-5 diagnostic criteria. We will compare the mean scores in each arm.
Daily functioning (WHODAS 2.0- 12-item version) | Baseline Assessment; Follow up at 12 weeks post-counselling (18 weeks after baseline); Follow up at 47 weeks post-counselling (53 weeks after baseline)
  The WHO Disability Assessment Schedule (WHODAS 2.0) a 12-items measure will be used to assess functional impairment across six domains of life over the past 30 days. These include cognition, mobility, self-care, getting along with people, life activities, and participation in society. The total score ranges between 0 to 48 and a higher score indicates a greater difficulty in functioning. We will compare the mean scores in each arm.
Modified Collective Self-Esteem Scale | Baseline Assessment; Follow up at 12 weeks post-counselling (18 weeks after baseline); Follow up at 47 weeks after PM+ counselling completion (53 weeks after baseline assessment).
  Modified Collective Self-Esteem Scale will be used to assess participants' attitudes, feelings, and perceptions related to their membership in the LGBTIQA+ community. This tool measures sense of personal worth within the group, public perceptions of the group, the importance of group membership to personal identity, and the individual's sense of contribution and belonging. The total score ranges from 16 to 112 and higher total scores indicate more positive collective self-esteem related to the sexual and gender minority group membership. We will compare the mean scores in each arm.
Neff's Self-Compassion Scale (Short- form) | Baseline Assessment; Follow up at 12 weeks post-counselling (18 weeks after baseline); Follow up at 47 weeks after PM+ counselling completion (53 weeks after baseline assessment).
  The Neff's Self-Compassion Scale (short form) will be used to assess participants' capacity for self-compassion, particularly how they respond to themselves during times of failure, difficulty, or emotional distress. This scale measures components such as self-kindness, self-judgement, common humanity, isolation and mindfulness. The total score ranges from 12 to 60 and a higher total score reflects greater self-compassion. We will compare the mean scores in each arm.
MOS Modified Social Support Survey- Five Item Version (MSSS-5) | Baseline Assessment; Follow up at 47 weeks post-counselling (53 weeks after baseline).
  The MOS Modified Social Support Survey will be used to assess participants' perceived social support. MSSS-5 includes five items that measures the availability of various types of support such as emotional/informational, tangible, affectionate, and positive social interaction. Participants rate each item on a 5-point Likert scale (1=none of the item, 5=all the time) reflecting the frequency of available support in the past 4 weeks. The total scores ranges from 5 to 25 with higher scores indicating greater perceived social support. We will compare the mean scores in each arm.
Modified Safety Planning Checklist | Baseline Assessment; Follow up at 12 weeks post-counselling (18 weeks after baseline); Follow up at 47 weeks after PM+ counselling completion (53 weeks after baseline assessment).
  Modified Safety Planning Checklist will be used to assess participants' use of personal safety strategies in response to potential violence. This tool covers practical activities such as securing a safe place to stay, keeping essential documents or things (e.g., certificates, medicines etc.), preparing an emergency safety plan, using safety codes with trusted contacts, and keeping contact to emergency communication and contact lists.
Use of Community Resources | Baseline Assessment; Follow up at 12 weeks post-counselling (18 weeks after baseline); Follow up at 47 weeks after PM+ counselling completion (53 weeks after baseline assessment).
  This tool will be used to measure participants' use of community-based services for violence prevention and support. It captures both formal and informal support systems utilized by the participants (yes vs. no) across different time periods (from the past month as baseline to the past 12 months at the last follow-up) and assesses their level of satisfaction rated on a 5-point Likert scale (1=Not satisfied at all, 5= Very satisfied) with each available local support service in the community.
Psychological Outcomes | Intervention arm: Pre-counseling, during sessions 2-5, Follow-up 1 at one-week post-counseling and Follow-up 2 at 12 weeks after post-counseling. Enhanced usual care arm: Baseline, Follow-up 1 at 7 weeks, and Follow-up 2 at 18 weeks post-baseline.
  The Psychological Outcomes Profile (PSYCHLOPS) is a participant-reported outcome measure to evaluate perceived psychological change over time. It consists of four items that assess problems, functioning, and overall well-being. Each item is rated on a 6-point ordinal scale (0-5), with a total score range of 0-20; higher scores indicate greater psychological distress. One additional item assesses suicidal ideation and is used solely for safety monitoring. Participants also provide narrative responses related to their current concerns, which will be analyzed qualitatively. The tool includes a post-intervention item assessing perceived change (rated from "feeling much better" to "feeling much worse"). Quantitative scores will be analyzed using mean change from baseline between study arms. Qualitative responses will be thematically analyzed to identify common themes and concerns.

OTHER OUTCOMES:
Perceived feasibility and acceptability of SAATHI intervention (Augmented PM+ Model) | This measure will be assessed before the trial begins and throughout the trial period, up to the final follow up (Follow up 3) at 47 weeks after post-counselling (53 weeks after baseline assessment).
  This outcome will focus on the following factors:
  1. Need of adapting PM+ and safety planning to the social and cultural context of sexual and gender minorities. Qualitative themes will be derived through analysis of data from interviews and focus group discussions.
  2. Perceptions of facilitators and barriers to implementation from the perspective of key stakeholders, including peer counselors, LGBTIQA+ participants, community leaders, NGO representatives, and healthcare professionals. Qualitative themes will be derived through analysis of data from interviews and focus group discussions.
  3. Participant retention rate in SAATHI intervention sessions. The unit of measure will be percentage scores derived from implementation fidelity checklist scores, session completion rates, and exit client interviews.
Process evaluation of SAATHI intervention (Augmented PM+ Model) | Process evaluation activities will be conducted throughout the intervention delivery period, and up to the final follow-up at 53 weeks after baseline assessment. Interim findings may be used to refine ongoing implementation.
  1. Adherence to the intervention manual and quality of counselling sessions which will be measured through session observations, documentation, and exit client interviews. The unit of measure will be percentage adherence scores.
  2. Experiences with contextual factors, mechanisms of impact, and sustainability of the peer-led SAATHI intervention. Qualitative themes will be derived through analysis of data from interviews and focus group discussions.
  3. Barriers and facilitators to implementation from participant and peer counselor perspectives. Qualitative themes will be derived through analysis of data from interviews.
Evaluation of Competency-Based Training for Peer Providers of the SAATHI intervention (Augmented PM+ Model) | This evaluation will be conducted both before and after the competency-based training of LGBTIQA+ peers.
  The training aims to enhance following areas:
  * Core competencies measured by the ENACT (ENhancing Assessment of Common Therapeutic factors) tool.
  * Delivery-specific competencies measured by the EQUIP PM+ competency rating scale.
  Peer advocate performance will be evaluated pre- and post-training using a standardized observation tool. This involves assessing behaviors during role plays. Each skill will be scored on a four-level scale: level 1 exhibits unhelpful or potentially harmful behavior; level 2 demonstrates no or only partial basic skills; level 3 demonstrates all basic helping skills; level 4 demonstrates all basic helping skills plus one or more advanced skills. The unit of measure will be competency levels scored using standardized tools. In addition, peer advocates' practice will be assessed through direct observations of real counselling sessions. In addition, in depth interviews will explore their experiences of applying the competencies in real-world settings.

CONTACTS AND LOCATIONS:
Locations (6):
- Nepal (6):
  - SAATHI Program Chitwan site, Chitwan, Bagmati
  - SAATHI Program Kathmandu and Lalitpur site, Kathmandu, Bagmati
  - SAATHI Program Makwanpur site, Makwanpur, Bagmati
  - SAATHI Program Dhanusha site, Dhanusha, Madhesh
  - SAATHI Program Parsa site, Parsa, Madhesh
  - SAATHI Program Sarlahi site, Sarlahi, Madhesh

IPD SHARING:
Plan to Share IPD: Yes
This study evaluates the effectiveness of a psychosocial intervention among a highly vulnerable and marginalized population-sexual and gender minorities-who experience daily abuse, discrimination, and marginalization in Nepalese society. The study collects sensitive data, including mental health status, exposure to violence, and related psychosocial factors.
  To protect participants privacy, a de-identified dataset will be shared only after the publication of findings related to primary and secondary outcomes. The shared dataset will exclude identifying variables such as age, study district, and gender identity.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2031-December 2031
Access Criteria: Collaborators and qualified independent researchers may request access to the de-identified individual participant data and supporting documentation (e.g., codebooks and analysis plan) by submitting reasonable written request to the principal investigator (PI). Contact information will be provided in the scientific publications associated with the study.